CLINICAL TRIAL: NCT04033744
Title: Prevention of Mandibular Third Molar Extraction- Associated Periodontal Defects Using Platelet-Rich Fibrin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Naples (Other)
Responsible Party: Principal Investigator, Gilberto Sammartino, Full Professor, University of Naples
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 56/15
Record Dates: First submitted 2019-07-22; First posted 2019-07-26 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-07

CONDITIONS: Periodontal; Lesion; Periodontal Pocket; Molar, Third
Keywords: Molar, Third; Platelet-Rich Fibrin
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: One clinician, not involved in patient treatment and not aware of what therapeutic approach was used for the different sites of treatment, performed all clinical measurements (PD, CAL, gingival recession, plaque index and gingival bleeding index) before and after 12 and 18 weeks of surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF (platelet-rich fibrin) (Experimental): PRF will be used after the extraction of the third molar to prevent periodontal defects to second molar
  Interventions: Procedure: extraction of mandibular third molar
- spontaneous healing (Active Comparator): after the extraction of the third molar the socket will be left to heal spontaneously
  Interventions: Procedure: extraction of mandibular third molar

INTERVENTIONS:
Procedure: extraction of mandibular third molar — After loco-regional anesthesia was administered, a full-thickness mucoperiosteal flap was raised. The flap incision was extended from the vestibular side of the retromolar trigon to the second molar, corresponding to its distolingual cusp. The incision continued intrasulcular at the second molar and proceeded with a release incision distally to the papilla between the first and second molars, on a 45° angle. An osteotomy using a Lindemann burr under constant irrigation, followed by an odontotomy using a diamond burr was performed, if necessary

SUMMARY:
The extraction of deep impacted mandibular third molar may cause periodontal defects at the distal root of the second molar. The aim of this study was to evaluate the ability of platelet-rich fibrin (PRF) in preventing periodontal complications at the distal root of the second molar adjacent to the extracted third molar.

DETAILED DESCRIPTION:
Eighteen young patients with bilateral impacted mandibular third molars will be selected. All 36 cases of impactions will be selected for a split mouth study and randomly treated by using 2 different therapeutic approaches, thereby yielding 2 different study groups, each of which is composed of 18 cases: in one side the post-extraction socket is left healing spontaneously, on the other side the socket is filled with PRF.

CAL at the distal surface of the lower second molar is chosen as primary outcome.

Criteria will be the presence of a pocket distal to the mandibular second molar with a probing depth >7 mm and a probing clinical attachment level >6mm.

This study was designed as a single-blind research since subjects will be unaware of their treatment allocation. A software will be used to produce a random sequence of 18 integer numbers without duplicates generated from atmospheric noise and concealed in closed envelopes by one of the investigators. At the time of the patient's first surgery, the envelope will be opened and patient allocated either to group 1 (PRF on the right side, spontaneous healing on the left side), for allocation numbers 1-9, or group 2 (spontaneous healing on the right side, PRF on the left side), for allocation numbers 10-18.

One clinician, not involved in patient treatment and not aware of what therapeutic approach used for the different sites of treatment, will perform all clinical measurements (PD, CAL, gingival recession, plaque index and gingival bleeding index) before and after 12 and 18 weeks of surgery.

Clinical and radiographical measurements will be recorded at 12 and 18 weeks after the surgery. The Student t test will be used to compare the differences between the 2 groups.

ELIGIBILITY:
Inclusion criteria Patients of both genders and any race, between 18 and 35 year-old

* Periodontally health patients and treated periodontally compromised patients
* Enrollment on a regular supportive periodontal therapy (SPT) program.
* Full-mouth plaque score (FMPS)< 25% at baseline;
* Full-mouth bleeding score (FMBS)< 25% at baseline;
* Patients having bilateral mesioangular impacted mandibular third molars with the presence of a pocket distally to the mandibular second molar with a probing depth (PD) ≥7 mm
* Intact buccal and lingual cortical bone of the post-extraction site

Exclusion Criteria:

* General contra-indications for surgery (systemic disease, compromised immune system etc);
* Tobacco smoking
* Pregnancy and lactation
* Untreated periodontal conditions;
* Acute infection in the site of the extraction
* Patients taking any medications which might interfere with coagulation
* Platelet count < 150000/mm3

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-07 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Clinical attachment level change | 12 and 18 weeks
  the clinical attachment level is the distance between the gingival margin to the cemento-enamel junction.
  the measurement is made by using a Williams periodontal probe. Differences in changes are measured from baseline to 12 and 18 weeks.

SECONDARY OUTCOMES:
probing depth change | 12 and 18 weeks
  The probing depth is the distance from the free end of the gingival margin to the bottom of the periodontal pocket. The measurement is made by using a Williams periodontal probe. Differences in changes are measured from baseline to 12 and 18 weeks.
gingival recession change | 12 and 18 weeks
  The distance between the cemento-enamel junction and gingival margin gives the level of recession.
  The measurement is made by using a Williams periodontal probe. Differences in changes are measured from baseline to 12 and 18 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto Sammartino, Professor, Principal Investigator — Federico II University
Locations (1):
- Gilberto Sammartino, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cabaro S, D'Esposito V, Gasparro R, Borriello F, Granata F, Mosca G, Passaretti F, Sammartino JC, Beguinot F, Sammartino G, Formisano P, Riccitiello F. White cell and platelet content affects the release of bioactive factors in different blood-derived scaffolds. Platelets. 2018 Jul;29(5):463-467. doi: 10.1080/09537104.2017.1319046. Epub 2017 Jun 21. PMID 28635382
- [Result] Sammartino G, Dohan Ehrenfest DM, Carile F, Tia M, Bucci P. Prevention of hemorrhagic complications after dental extractions into open heart surgery patients under anticoagulant therapy: the use of leukocyte- and platelet-rich fibrin. J Oral Implantol. 2011 Dec;37(6):681-90. doi: 10.1563/AAID-JOI-D-11-00001. Epub 2011 Jun 30. PMID 21718187
- [Result] Sammartino G, Tia M, Marenzi G, di Lauro AE, D'Agostino E, Claudio PP. Use of autologous platelet-rich plasma (PRP) in periodontal defect treatment after extraction of impacted mandibular third molars. J Oral Maxillofac Surg. 2005 Jun;63(6):766-70. doi: 10.1016/j.joms.2005.02.010. PMID 15944972